CLINICAL TRIAL: NCT02718014
Title: Evaluation of Periodontal Response to Non Surgical Therapy in Pre and Post Menopausal Women With Periodontitis
Acronym: EPRNPPMP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, J S Prasanna, DR, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PMVIDSRC
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Periodontitis; Menopause; Plaque; Inflammation
Keywords: Non Surgical Therapy
MeSH Terms: conditions — Periodontitis; Plaque, Amyloid; Inflammation | interventions — Tooth Exfoliation; Root Planing; Urocortins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pre menopause with periodontitis (Other): non surgical periodontal therapy (SCALING & ROOT PLANING) (SRP)
  Interventions: Other: scaling and root planing (srp)
- post menopause with periodontitis (Other): non surgical periodontal therapy (SCALING & ROOT PLANING) (SRP)
  Interventions: Other: scaling and root planing (srp)

INTERVENTIONS:
Other: scaling and root planing (srp)

SUMMARY:
The present study was evaluated periodontal status in pre and post-menopausal women with periodontitis following non-surgical therapy.

DETAILED DESCRIPTION:
AIM: The aim of the present study was to evaluate periodontal status in pre and post-menopausal women with periodontitis following non-surgical therapy.

MATERIALS AND METHODS: Periodontal status was measured by Periodontal index (PRI), and oral hygiene status was measured by plaque index (PI). Both the parameters were measured at baseline i.e before Scaling and Root Planing (SRP) and after 3 months intervals post treatment. SRP was done in both pre&post menopause groups.

ELIGIBILITY:
Inclusion Criteria:Patients should have at least 15 natural teeth remaining

* Non smokers
* Systemically healthy from past 6 months

Exclusion Criteria:Present or past smokers

* Below 40 years of age
* With gross oral pathology or tumors
* Patients on long term steroid medication
* Undergoing Hormone replacement therapy (HRT)
* Pregnant women or planning for pregnancy
* Those who have received periodontal therapy in the preceding 6 months
* Those that are under medication in the preceding 6 months
* Any systemic disorders or any medication that affects the periodontal status was excluded from this study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of periodontal response to non surgical therapy in pre and post menopausal women with periodontitis | 3 months
  pocket depth reduction calculated with PRI index
Evaluation of periodontal response to non surgical therapy in pre and post menopausal | 3 months
  plaque scores was calculated with Silness and Loe index

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buencamino MC, Palomo L, Thacker HL. How menopause affects oral health, and what we can do about it. Cleve Clin J Med. 2009 Aug;76(8):467-75. doi: 10.3949/ccjm.76a.08095. PMID 19652040
- [Background] Deasy MJ, Vogel RI. Female sex hormonal factors in periodontal disease. Ann Dent. 1976 Fall;35(3):42-6. PMID 788632
- [Background] Aznar Reig A, Zamora Madarias E, Bonilla Mir F, Lopez Campos J, Majua Delgado R. [Hepatic satelite lesion in biliary calculi]. Rev Esp Enferm Apar Dig. 1968 Aug-Sep;27(7):1019-40. No abstract available. Spanish. PMID 4195183
- [Result] Yobs AR, Plott AE, Hicklin MD, Coleman SA, Johnston WW, Ashton PR, Rube IF, Watts JC, Naib ZM, Wood RJ, et al. Retrospective evaluation of gynecologic cytodiagnosis. II. Interlaboratory reproducibility as shown in rescreening large consecutive samples of reported cases. Acta Cytol. 1987 Nov-Dec;31(6):900-10. PMID 3425152
- [Result] Tobin JO, Watkins ID, Woodhead S, Mitchell RG. Epidemiological studies using monoclonal antibodies to Legionella pneumophila serogroup 1. Isr J Med Sci. 1986 Oct;22(10):711-4. PMID 3793432